CLINICAL TRIAL: NCT01699815
Title: Time of Intravenous Acetaminophen Administration for Total Hip Arthroplasty
Brief Title: Time of Intravenous Acetaminophen Administration
Acronym: TIAA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00036568
Record Dates: First submitted 2012-09-28; First posted 2012-10-04 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Osteoarthritis
Keywords: acetaminophen; timing; arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preemptive group (Active Comparator): The preemptive group will receive one dose of 1 gram of IV acetaminophen every 6 hours x 24 hours with the first dose administered within 60 minutes prior to incision. Each infusion will be administered over 15 minutes as recommended by manufacturer package insert.
  Interventions: Drug: Acetaminophen
- Closure group (Active Comparator): The closure group will receive one dose of 1 gram of IV acetaminophen every 6 hours x 24 hours with the first dose administered upon onset of skin closure.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen

SUMMARY:
The purpose of the study is to examine the effects of timing of administration of intravenous (IV) acetaminophen and how timing relates to analgesic efficacy as measured by postoperative pain scores. A maximum of 138 patients meeting inclusion criteria who present for a scheduled total hip replacement under general anesthesia will be randomized into one of two arms: 1) the pre-closure group will receive the first dose administered upon onset of skin closure, 2) the preemptive group will receive the first dose administered within 60 minutes prior to incision. Both groups will receive subsequent doses every 6 hours x 24 hours.

DETAILED DESCRIPTION:
The purpose of the study is to examine the effects of timing of administration of intravenous (IV) acetaminophen and how timing relates to analgesic efficacy as measured by postoperative pain scores. A maximum of 138 patients meeting inclusion criteria who present for a scheduled total hip replacement under general anesthesia will be randomized into one of two arms: 1) the closure group will receive the first dose of one gram of intravenous acetaminophen administered upon onset of skin closure, 2) the preemptive group will receive the first dose of one gram of intravenous acetaminophen administered within 60 minutes prior to incision. Both groups will receive subsequent doses of one gram of intravenous acetaminophen every 6 hours x 24 hours. The maximum dose in a 24 hour period will not exceed 4 grams according to FDA recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients 30-75 years of age weighing ≥55 kg scheduled for elective total hip arthroplasty performed under general anesthesia will be included. As determined by the anesthesia team assigned to the case, eligible patients will also be assigned ASA physical status of I, II, or III and deemed capable of reporting their perceived pain using numeric pain scales and capable of operating a patient controlled anesthesia (PCA) device.

Exclusion Criteria:

* Exclusion criteria include known allergy, hypersensitivity, or contraindication to acetaminophen, history of alcohol or drug abuse, prisoners, emergency THAs, patients with chronic malnutrition or a body mass index (BMI) < 18 kg/m2 and non-English speaking patients. Additional exclusion criteria include impaired liver function defined as AST and ALT each ≥ twice normal limits and renal dysfunction (creatinine >2.0 mg/dl).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia C Muckler, DNP, Principal Investigator — Duke Health
Locations (1):
- Durham Regional Hospital, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Preemptive Group: The preemptive group will receive one dose of 1 gram of IV acetaminophen every 6 hours x 24 hours with the first dose administered within 60 minutes prior to incision. Each infusion will be administered over 15 minutes as recommended by manufacturer package insert.
  Acetaminophen
- Closure Group: The closure group will receive one dose of 1 gram of IV acetaminophen every 6 hours x 24 hours with the first dose administered upon onset of skin closure.
  Acetaminophen
Period: Overall Study
Arm/Group | Preemptive Group | Closure Group
Started | 62 | 64
Completed | 57 | 56
Not Completed | 5 | 8
Not completed — Protocol Violation | 4 | 7
Not completed — record could not be located | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preemptive Group | Closure Group | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Full Range); unit: years] | 60.5 [37 to 74] | 61.7 [35 to 75] | 61.1 [35 to 75]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 56 | 113
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 18 | 50
  Male | 25 | 38 | 63
Region of Enrollment [Number; unit: participants]
  United States | 57 | 56 | 113

OUTCOME MEASURES:

1. Primary Outcome: Changes in Postoperative Pain Scores
Description: To compare analgesic efficacy as measured by changes in postoperative pain scores assessed preoperatively, at 6, 12, 18, and 24 hours following the initial administration of the study drug. Pain scores are assessed on a scale of 0 - 10. 0 = No Pain; 10 = Worst Possible Pain
Time Frame: preoperatively (baseline), post-anesthesia care unit (PACU or recovery room) arrival (2-3 hour), and 6,12, 18, and 24 hours following the initial administration of the study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preemptive Group | Closure Group
Number analyzed (Participants) | 57 | 56
units on a scale
  preoperatively (baseline) | 2.7 (1.41) | 2.5 (2.69)
  PACU arrival (2-3 hour) | 0.9 (2.3) | 1.5 (3.1)
  6 hrs post study drug | 2.6 (2.75) | 2.6 (2.21)
  12 hrs post study drug | 2.5 (2.69) | 2.3 (2.05)
  18 hrs post study drug | 2.7 (2.45) | 2.6 (2.28)
  24 hrs post study drug | 3.0 (2.53) | 2.9 (2.44)

2. Secondary Outcome: Pain Medication Consumption Rates
Description: Number of participants who required rescue pain medication. Rescue pain medications is defined as administration of pain medication in excess of standard postoperative pain medication orders.
Time Frame: Arrival to post-anesthesia care unit (PACU or recovery room) (2-3 hours post baseline) to 24 hours post administration of study drug
Measure: Number; unit: participants
Arm/Group | Preemptive Group | Closure Group
Number analyzed (Participants) | 57 | 56
participants | 50 | 42

3. Other Pre Specified Outcome: Average Length of Stay (LOS)
Description: To compare patient length of stay (LOS) between groups as measured by day of discharge minus day of admission.
Time Frame: Baseline to discharge (1-4 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Preemptive Group | Closure Group
Number analyzed (Participants) | 57 | 56
days | 2.5 (0.5) | 2.0 (0)

ADVERSE EVENTS:
Groups:
- Preemptive Group: The preemptive group will receive one dose of 1 gram of IV acetaminophen every 6 hours x 24 hours with the first dose administered within 60 minutes prior to incision. Each infusion will be administered over 15 minutes as recommended for OfirmevTM administration.
  Acetaminophen
Arm/Group | Preemptive Group | Closure Group
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 0/57 | 1/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preemptive Group (N=57) | Closure Group (N=56)
Seizure (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No